CLINICAL TRIAL: NCT01515761
Title: POsition of Leads in Advanced heaRt Failure: the POLAR Study - A 6 Month, Observational, Mult-centered, Blinded, Randomized Study to Determine if Lead Positioning in the Lateral Wall of LV in Patients Meeting Criteria for CRT Plays a Role in Determining Myocardial Function and Affect the Severity of Mitral Regurgitation
Brief Title: POsition of Leads in Advanced heaRt Failure: the POLAR Study
Acronym: POLAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sergio Thal, M.D. (U.S. Federal Agency)
Collaborators: Medtronic (Industry); Lexington VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Sergio Thal, M.D., Electrophyisology Laboratory Director, Southern Arizona VA Health Care System
Organization: Southern Arizona VA Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PIIT1A
Record Dates: First submitted 2012-01-12; First posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Cardiac Resynchronization Therapy; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Postero-lateral (Active Comparator): Left ventricular lateral wall lead position
  Interventions: Procedure: Postero-lateral
- Antero-lateral (Active Comparator): Left ventricular lateral wall lead position
  Interventions: Procedure: Antero-Lateral

INTERVENTIONS:
Procedure: Postero-lateral — A device implant procedure will be performed under the standard of care technique with the right ventricular lead at the right ventricular apex and the left ventricular lead targeting or postero-lateral area of the LV based on pre-procedure randomization.
  Arms: Postero-lateral
Procedure: Antero-Lateral — A device implant procedure will be performed under the standard of care technique with the right ventricular lead at the right ventricular apex and the left ventricular lead targeting or antero-lateral area of the LV based on pre-procedure randomization.
  Arms: Antero-lateral

SUMMARY:
The primary objective is to determine if lead positioning in the lateral wall of the left ventricle in patients meeting criteria for cardiac resynchronization therapy plays a role in determining myocardial function and affects the severity of mitral regurgitation.

DETAILED DESCRIPTION:
This is a 6 month, multi-centered, blinded, randomized study. Approximately 60 patients will join this study. Two groups, based on lead position, will be studied with thirty (30) patients randomized into each group.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets the general indications for an implantable cardioverter defibrillator (ICD) with LV systolic function ≤ 35% as defined by echocardiography.
* Subject has moderate or severe heart failure, defined as NYHA Class III-IV for at least 90 days prior to enrollment.
* Subject has optimal pharmacological heart failure therapy for at least 30 days prior to enrollment.
* Subject has a 12-lead electrocardiogram (ECG) obtained no more than 90 days prior to enrollment documenting a sinus rate > 50 bpm and PR interval < 320 ms measured from any two leads.
* 12 lead ECG with left bundle brunch block morphology and a QRS duration of at least 120 msec.
* Subject has creatinine < 2.5 mg/dL obtained no more than 30 days prior to enrollment.
* Subject has left ventricular ejection fraction < 35% by echocardiogram no more than 1 year prior to enrollment.
* Subject is willing and capable of undergoing a device implant and participating in all testing associated with this clinical investigation.
* Subject has a life expectancy of more than 180 days, per physician discretion.
* Subject is age 18 or above, or of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

* Subject has right bundle branch block morphology on a 12-lead ECG obtained no more than 90 days prior to enrollment.
* Subject had previous cardiac resynchronization therapy, a previous coronary venous lead, or meets the general indications for anti-bradycardia pacing defined as ventricular pacing > 40% by pacemaker interrogation.
* Subject has a neuromuscular, orthopedic, or other non-cardiac condition that prevents normal, unsupported walking.
* Subject has an atrial tachyarrhythmia that is permanent (i.e., does not terminate spontaneously and cannot be terminated with medical intervention) or persistent (i.e., can be terminated with medical intervention, but does not terminate spontaneously) within 30 days prior to enrollment.
* Subject currently requires dialysis.
* Subject has severe chronic obstructive pulmonary disease (COPD), defined as FEV1/FVC < 60%, or as defined by a physician.
* Subject has had a myocardial infarction within 30 days prior to enrollment or coronary artery disease (CAD) in which surgical or percutaneous correction was performed within 30 days prior to enrollment.
* Subject has hypertrophic obstructive cardiomyopathy or infiltrative cardiomyopathy (e.g., amyloidosis, sarcoidosis).
* Subject is on IV inotropic agents.
* Subject has any mitral valve prosthesis, or a mechanical aortic or tricuspid prosthesis
* Subject is enrolled in any concurrent study, without Medtronic written approval, which may confound the results of this study.
* Subject is pregnant or planning to get pregnant.
* Subject requires oxygen for medical reasons other than CHF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Change (reduction) in left ventricular end systolic volume (LVESV) | 3 and 6 months
Change in 6 minute walk tests | 6 weeks, 3 and 6 months

SECONDARY OUTCOMES:
Myocardial performance as measured by myocardial performance index (MPI) | 6 months
Papillary muscle velocity as determined by tissue doppler | 6 months
Progression of mitral regurgitation | 6 months
  as measured by regurgitant volume, mitral regurgitation fraction and effective regurgitant orifice area
Minnesota living heart failure survey | 6 weeks, 3 and 6 months
Chronic heart failure hospitalizations | Monitored during study participation ~ 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Thal, M.D., Principal Investigator — Southern Arizona VA Health Care System
Locations (2):
- United States (2):
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Lexington VA Medical Center, Lexington, Kentucky